CLINICAL TRIAL: NCT01521403
Title: Is it Effective to Treat Patients With Blastocystis Hominis Infection? A Double-blind Placebo Controlled Randomized Trial
Brief Title: Is it Effective to Treat Patients With Blastocystis Hominis Infection?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Serge de Valliere, MD, MSc, Consultant, Principal Investigator, University of Lausanne Hospitals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVMV-Blastocystis hominis
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Blastocystis Hominis Infections
Keywords: Blastocystis hominis; Metronidazole
MeSH Terms: conditions — Blastocystis Infections | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole (Active Comparator): Metronidazole 3x500 mg per day for 10 days
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Placebo 3x1 tablet per day for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metronidazole — 3x500 mg/day for 10 days
  Arms: Metronidazole
Drug: Placebo — 3x1 tablet per day for 10 days
  Arms: Placebo

SUMMARY:
The objective of this study is to determine whether in the setting of primary health care it is effective to treat with metronidazole returning travellers with gastrointestinal symptoms and B. hominis in the stool or not.

DETAILED DESCRIPTION:
Prevalence of B. hominis is between 30-50% in developing countries. Many travellers visit developing countries and are therefore at risk to be infected by this parasite. It's frequent that travellers return from developing countries with gastro-intestinal symptoms and approximately 10% of them have B. hominis as the sole parasite identified in the stools. Some anti-infective drugs, including metronidazole, trimethoprim-sulfamethoxazole and nitazoxanide, have shown to have activity against B. hominis, but there is still controversy about the pathogenic potential of B. hominis and there is no consensus about the indications for treatment.

It is hypothesised that metronidazole is more effective than placebo in returning travellers with gastrointestinal symptoms and B. hominis as the sole intestinal parasite identified in the stool.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Gastrointestinal symptoms for more than 10 days
* B. hominis in any quantity in at least one stool specimen out of 3 examined
* No other pathogenic micro-organism identified

Exclusion Criteria:

* Fever > 37.5°
* bloody diarrhoea
* weight loss > 10% of usual body weight
* significant decrease of general condition
* oncological diseases
* immune deficiencies
* known chronic intestinal diseases
* use of anti-protozoan drugs in the last 2 weeks
* use of anti-coagulant treatment or antabuse
* pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-11 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of gastro-intestinal symptoms | 10-14 days after treatment with Metronidazol
  The improvement of the following symptoms will be evaluated:
  * Presence of unusually soft or unformed stools in the last 3 days (yes or no)
  * Average number of stools per day in the last 3 days
  * Maximal abdominal pain in the last 3 days on a scale from 0-10
  * Bloating in last 3 days on a scale from 0-10
  * Flatulence in last 3 days on a scale from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Serge de Valliere, MD, MSc, Principal Investigator — Travel Clinic, Department of Ambulatory Care and Community Medicine, University Hospital of Lausanne, Switzerland
Locations (1):
- Travel Clinic, Department of Ambulatory Care and Community Medicine, University Hospital of Lausanne, Switzerland, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No